CLINICAL TRIAL: NCT02285764
Title: NIGO Health- Nutritional Intervention During Gestation and Offspring Health
Brief Title: Nutritional Intervention During Gestation and Offspring Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AL10
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Maternal Glycemia
MeSH Terms: interventions — Dietary Supplements; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional Supplement (Experimental): One 237 ml oral supplement consumed two times a day; Not commercially available.
  Interventions: Other: Nutritional Supplement
- Standard of Care (Other): As determined by the study site
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Nutritional Supplement — Modified carbohydrate
  Arms: Nutritional Supplement
Other: Standard of Care — As determined by the study site
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to investigate the potential effects of a modified carbohydrate nutritional product for obese pregnant women to reduce maternal glycemia.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated an ICF, approved by an IEC/IRB and provided applicable privacy authorization prior to any participation in the study.
* Obese (BMI ≥ 30) as determined by pre-pregnancy BMI.
* ≥18 years of age.
* ≥15+0 but ≤16+6 weeks gestation with a singleton pregnancy.
* Willing to follow supplementation protocol and follow appropriate nutritional guidance and refrain from consuming other caloric nutritional supplements that are not approved by the study staff, if applicable.
* Willing to provide body composition measures on infant at birth.
* Willing to consider additional measures if follow-up studies are conducted.

Exclusion Criteria:

* Adverse maternal and/or fetal medical history which is expected to alter blood glucose regulations.
* Previously diagnosed diabetes, previous gestational diabetes, systemic lupus erythematodes, anti-phospholipid syndrome, known renal disease, treated hypertension, uncontrolled hypothyroidism and/or cancer.
* Taking medications that can impact blood glucose.
* Previous bariatric surgery.
* Lactose intolerant and/or has milk protein allergy or requires a special diet regime.
* Participating in another clinical trial that would impact participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Maternal Oral Glucose Tolerance Test (OGTT) | 27-28 weeks gestation
  2 hour OGTT

SECONDARY OUTCOMES:
Neonatal Body Composition | Birth - 72 hours
Maternal Fasting Blood Glucose | 34-36 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Elena Oliveros Delgado, BSc, MSc, Study Chair — Abbott Nutrition; Ricardo Rueda, MD, PhD, Study Chair — Abbott Nutrition
Locations (3):
- Ludwig-Maximilians-University of Munich, Dr. von Hauner Children's Hospital, München, Germany
- Spain (2):
  - University of Granda, Granada
  - University Clinical Hospital San Cecilio, Granada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] G Bermudez M, Garcia-Ricobaraza M, Garcia-Santos JA, Segura MT, Puertas-Prieto A, Gallo-Vallejo JL, Padilla-Vinuesa C, Koletzko B, Baggs GE, Oliveros E, Rueda R, Campoy C. Effect of a Low Glycemic Index/Slow Digesting (LGI/SD) Carbohydrate Product on Maternal Glycemia and Neonatal Body Composition in Obese Pregnant Women: The NIGOHealth Randomized Clinical Trial. Nutrients. 2025 Jun 5;17(11):1942. doi: 10.3390/nu17111942. PMID 40507210